CLINICAL TRIAL: NCT06723587
Title: Chronic Effects of the Use of Instep Weights on Technical, Physical and Perceptual Parameters in Young Male Soccer Players
Brief Title: Chronic Effects of the Use of Instep Weights on Specific Capacities in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RCTPI001
Record Dates: First submitted 2024-12-02; First posted 2024-12-09 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Soccer; Physical Stress; Physical Performance
Keywords: Performance; Accuracy; Agility; Soccer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instep weights (Experimental): Instep weight use
  Interventions: Other: Instep weights use
- No instep weights (No Intervention): No instep weight.

INTERVENTIONS:
Other: Instep weights use — Players will perform their scheduled training sessions while wearing a 150-gram instep weight. The use of instep weights in the intervention group will be introduced progressively and gradually, increasing both the frequency of sessions and the duration of their use.
  During weeks 1-2, instep weights will be used in one training session per week. During weeks 3-5, will be used in two training sessions per week.
  And during weeks 6-8, will be used in three training sessions per week.
  The duration of instep weight usage within each session will increase by 5% weekly, starting at 40% in Week 1 and reaching 75% by Week 8.
  Arms: Instep weights

SUMMARY:
The main goal of this randomized controlled trial (RCT) is to evaluate the chronic effects of using instep weights on technical, physical (conditional), and perceptual parameters in amateur male soccer players.

The secondary objective will be to propose a training methodology using instep weights to enhance athletic performance.

The following hypotheses are formulated based on the objectives outlined previously.

Hypothesis 1: the use of instep weights will enhance performance in ball striking speed, change of direction ability, and repeated sprint capacity.

Hypothesis 2: the use of instep weights will negatively affect performance in ball striking accuracy and ball control.

Hypothesis 3: the use of instep weights will not produce adverse effects on perceived exertion, groin pain or reduce maximal adductor, quadriceps and hamstring muscle contraction values.

DETAILED DESCRIPTION:
A RCT will be performed and players will be randomly assigned in one of the two groups (experimental or control).

Players will attend their regular training sessions and the protocol will be divided into two phases:

* Phase 1: familiarization On the recruitment day, players will be briefed on the study procedures, followed by the reading and signing of informed consent forms. Familiarization with the study procedures will take place over the two weeks prior to the intervention phase. During this period, participants will practice all testing protocols once a week and will wear 100-gram instep weights in different training sessions.
* Phase 2: intervention During the intervention phase, all players who meet the inclusion and exclusion criteria will be recruited and will be randomly allocated into an intervention group (experimental) or a non-intervention group (control group). Randomization will be conducted by an external researcher using blocked randomization via a web-based tool (Urbinak, 1997). Both groups will undergo distinct interventions over an 8-week period.

The study will be conducted during the competitive season on artificial turf field under consistent environmental conditions. Players will wear soccer boots for all testing procedures. Testing will occur at three time points:

* Pre-intervention: first day of Week 1 to collect baseline data.
* Mid-intervention: first day of Week 5.
* Post-intervention: first day of Week 9.

ELIGIBILITY:
Inclusion Criteria:

* amateur young male soccer player (under federation regulation)
* minimum three years of experience playing soccer
* train 3 days/week and 5 hours/week (minimum)

Exclusion Criteria:

* Injured players
* Goalkeepers
* Players unable to perform at their best
* Players that will miss more than two training sessions
* Players under medication or using performance enhancement supplements
* Players under 16 years old

Ages: 16 Years to 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Hip and Groin Outcome Score (HAGOS) | Pre-intervention (first day of week 1), mid-intervention (first day of week 5), and post-intervention (first day of week 9)
  The HAGOS was first described and validated in 2011 in the British Journal of Sports Medicine (Thorborg et al., 2011). It reliably assesses a patient's perception of disability, discomfort, or issues related to the hip and/or groin region. In addition to perceived dysfunction, the questionnaire also measures actual disability. HAGOS was designed to evaluate both short-term functional changes, such as those observed week-to-week during therapy, and long-term outcomes, such as the natural progression of a condition.
  HAGOS consists of six subscales scored from 0 (extreme) to 100 (no existance) hip/groin problems. Scales evaluate: Symptoms; Pain ; Physical Function in Daily Living; Function in Sports and Recreation; Participation in Physical Activities and Quality of Life. With: 7, 10, 5, 8, 2 and 5 items for each subscale respectively.
  The final measure is a composite outcome measure obtained by summing the values of the 6 subscales
Subjective perceptual well-being questionnaire measures change: RPE | The questionnaire will be administered within the first 15-20 minutes following the conclusion of each training session.
  Rate of Perceived Exertion (RPE) using the Borg (Borg, 1982) 0-10 scale (being 0 no exertion and 10 maximal exertion) will also be recorded. Players will respond one simple question: How hard was your session? Each player will complete the 0-to-10 scale without the presence of other players and will not see the values of other participants. Players will be allowed to mark a plus sign (interpreted as 0.5 point) alongside the integer value
Ball Striking Accuracy Test | Pre-intervention (first day of week 1), mid-intervention (first day of week 5), and post-intervention (first day of week 9)
  A precision screen (Nagasawa et al., 2011) measuring 7.3 meters wide by 2.4 meters high will be used to delineate target zones on a regulation football goal. The screen will have four openings (target zones) located in the top corners (Zones A and B) and bottom corners (Zones C and D). Each opening measures 1.5 meters wide by 0.8 meters high. Players will perform two strikes for each target zone in the following sequence: A, B, C, D. Accuracy will be assessed manually. A strike will score a point if the ball passes through the designated opening. Each successful strike scores one point, with a maximum total score of eight points (two successful strikes per zone). Accuracy will also be analyzed by high zones (A and B), low zones (C and D), and individual zones.
  Participants will be instructed to strike the ball with maximum power and precision.
  Official match balls used by the team for training and competition will be utilized, inflated to a pressure of 0.6-0.8 bar.
Ball Striking Velocity Test | Pre-intervention (first day of week 1), mid-intervention (first day of week 5), and post-intervention (first day of week 9)
  A Radar Stalker ATS II (Stalker®, USA) will be used to record ball velocity. Offering a time precision of 0.01 seconds, a velocity range of 1-1432.3 km/h, and the ability to detect ball motion up to 152.40 meters. Measurements will record the ball's speed in meters per second (m/s) as validated by previous studies (Ferraz et al., 2012; Tomas et al., 2014). The radar will be positioned directly behind the goal, 15 meters from the ball. The striking point will be at the penalty spot, 11 meters from the goal line.
  Participants will be instructed to strike the ball with maximum power and precision. Immediate feedback on velocity will be provided after each strike to encourage performance consistency or improvement.
  Official match balls used by the team for training and competition will be utilized, inflated to a pressure of 0.6-0.8 bar.
  Velocity data will be recorded (km/h) automatically by the radar.
Change of Direction (COD) and Ball Control | Pre-intervention (first day of week 1), mid-intervention (first day of week 5), and post-intervention (first day of week 9)
  The test evaluates the player's ability to change direction quickly and efficiently, as well as to control the ball while doing so. To evaluate these variables, the modified Barrow test (Bidaurrazaga et al., 2015) will be used.
  Players will start the test by positioning the foot they use most efficiently to begin the sprint at the starting point. They will then begin the test voluntarily, without waiting for a starting signal. The test will be performed in two conditions: without a ball and with a ball. Each player will perform the test twice in each condition, and the average result will be recorded. Results will be recorded using ChronoJump Boscosystem® photogates (Barcelona, Spain), with timing measurements conducted using Chronopic and recorded through Chronojump software version 2.2.1.
  Players will complete the test two times without the ball and two times with the ball, with a 2-minute rest between each attempt. The average values (sec) will be considered and analyzed.
Repeated Sprint Ability (RSA) | Pre-intervention (first day of week 1), mid-intervention (first day of week 5), and post-intervention (first day of week 9)
  To replicate the extreme demands of competition in terms of the number, duration, and recovery of sprints, a valid and reliable test (Aziz et al., 2008; Gabbett, 2010) will be used. This test aims to assess the ability of players to repeatedly perform high-intensity sprints with minimal recovery, reflecting the demands placed on athletes during competition.
  The test will consist of 6-8 sprints of 20 meters each, performed at maximal effort, with 20-second cycles between sprints. After each sprint, players will perform a 10-meter decelerationfollowed by a 10-meter active recovery (jogging). Results will be recorded using ChronoJump Boscosystem® photogates(Barcelona, Spain). The time measurements will be taken using Chronopic and recorded through Chronojump software version 2.2.1.
  The average values (sec) will be considered and analyzed.
Adductors Maximum Voluntary Contraction (MVC) | Pre-intervention (first day of week 1), mid-intervention (first day of week 5), and post-intervention (first day of week 9)
  MVC test will be used to assess the maximum force exerted by the hip adductors.
  A Lafayette Manual Muscle Testing System(Lafayette Instrument Company, Lafayette IN, USA) will be used to measure the muscle force.
  Two different procedures will be used to test the hip adductors(Esteve et al., 2018):
  1. Short Lever Test: resistance will be placed between the knees while the feet are positioned on the examination table. The hip will be in 45-degree flexion.
  2. Long Lever Test: resistance will be placed between the ankles, with the hip in neutral position (0° flexion).
  The maximum isometric force (Newtons;N) will be recorded as the average value of three attempts. For the hip adductor tests, both body mass and the length of the short and long levers (distance in cm between the body's center of mass and the point of resistance) will be measured for each player. Force values will then be normalized based on body weight and lever lengths and reported as N·m/kg.
Knee extensors Maximum Voluntary Contraction (MVC) | Pre-intervention (first day of week 1), mid-intervention (first day of week 5), and post-intervention (first day of week 9)
  The MVC test will be used to assess the maximum force exerted by the quadriceps. This is a valid and reliable test for evaluating the force capacity of the knee extensors (Alshahrani et al., 2023; Mentiplay et al., 2015).
  A Lafayette Manual Muscle Testing System(Lafayette Instrument Company, Lafayette IN, USA) will be used to measure the muscle force.
  To assess the quadriceps (knee extensors), the participant will be seated with the hips and knees flexed at 90°. The dynamometer will be placed on the anterior aspect of the lower leg, just proximal to the ankle joint (Alshahrani et al., 2023; Mentiplay et al., 2015).
  The maximum isometric force (measured in Newtons, N) will be recorded as the average value of three attempts.
  For the quadriceps test, the average force (N) from the three attempts will be normalized by body mass (measured in N/kg).
Knee flexors Maximum Voluntary Contraction (MVC) | Pre-intervention (first day of week 1), mid-intervention (first day of week 5), and post-intervention (first day of week 9)
  The MVC test will be used to assess the maximum force exerted by the hamstrings. This is a valid and reliable test for evaluating the force capacity of the knee flexors (Alshahrani et al., 2023; Mentiplay et al., 2015).
  A Lafayette Manual Muscle Testing System(Lafayette Instrument Company, Lafayette IN, USA) will be used to measure the muscle force.
  To assess the hamstrings (knee flexors), the participant will also be seated with the hips and knees flexed at 90°. The dynamometer will be positioned on the posterior aspect of the lower leg, proximal to the ankle joint (Alshahrani et al., 2023; Mentiplay et al., 2015).
  The maximum isometric force (measured in Newtons, N) will be recorded as the average value of three attempts.
  For the hamstring test, the average force (N) from the three attempts will be normalized by body mass (measured in N/kg).
Body mass | Pre-intervention (first day of week 1), mid-intervention (first day of week 5), and post-intervention (first day of week 9)
  Players body mass in kg will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Albert Altarriba-Bartes, PhD, Principal Investigator — Lecturer and Researcher
Locations (1):
- University of Vic-Central University of Catalonia, Vic, Spain

REFERENCES:
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Bidaurrazaga, I., Moreira, H., Lekue, J. A., Badiola, A., Figueiredo, A. J., & María, S. (2015). Applicability of an agility test in young players in the soccer field. Revista Brasileira de Medicina do Esporte, 21(2), 133-138.
- [Background] Aziz AR, Mukherjee S, Chia MY, Teh KC. Validity of the running repeated sprint ability test among playing positions and level of competitiveness in trained soccer players. Int J Sports Med. 2008 Oct;29(10):833-8. doi: 10.1055/s-2008-1038410. Epub 2008 Apr 9. PMID 18401804
- [Background] Esteve E, Rathleff MS, Vicens-Bordas J, Clausen MB, Holmich P, Sala L, Thorborg K. Preseason Adductor Squeeze Strength in 303 Spanish Male Soccer Athletes: A Cross-sectional Study. Orthop J Sports Med. 2018 Jan 11;6(1):2325967117747275. doi: 10.1177/2325967117747275. eCollection 2018 Jan. PMID 29349093
- [Background] Alshahrani MS, Reddy RS. Quadriceps Strength, Postural Stability, and Pain Mediation in Bilateral Knee Osteoarthritis: A Comparative Analysis with Healthy Controls. Diagnostics (Basel). 2023 Oct 1;13(19):3110. doi: 10.3390/diagnostics13193110. PMID 37835853
- [Background] Ferraz R, van den Tillaar R, Marques MC. The effect of fatigue on kicking velocity in soccer players. J Hum Kinet. 2012 Dec;35:97-107. doi: 10.2478/v10078-012-0083-8. Epub 2012 Dec 30. PMID 23486374
- [Background] Gabbett TJ. The development of a test of repeated-sprint ability for elite women's soccer players. J Strength Cond Res. 2010 May;24(5):1191-4. doi: 10.1519/JSC.0b013e3181d1568c. PMID 20386127
- [Background] Mentiplay BF, Perraton LG, Bower KJ, Adair B, Pua YH, Williams GP, McGaw R, Clark RA. Assessment of Lower Limb Muscle Strength and Power Using Hand-Held and Fixed Dynamometry: A Reliability and Validity Study. PLoS One. 2015 Oct 28;10(10):e0140822. doi: 10.1371/journal.pone.0140822. eCollection 2015. PMID 26509265
- [Background] Nagasawa, Y., Demura, S., Matsuda, S., Uchida, Y., & Demura, T. (2011). Effect of differences in kicking legs, kick directions, and kick skill on kicking accuracy in soccer players. Journal of Quantitative Analysis in Sports, 7(4), 9.
- [Background] Thorborg K, Holmich P, Christensen R, Petersen J, Roos EM. The Copenhagen Hip and Groin Outcome Score (HAGOS): development and validation according to the COSMIN checklist. Br J Sports Med. 2011 May;45(6):478-91. doi: 10.1136/bjsm.2010.080937. PMID 21478502
- [Background] Tomas M, Frantisek Z, Lucia M, Jaroslav T. Profile, correlation and structure of speed in youth elite soccer players. J Hum Kinet. 2014 Apr 9;40:149-59. doi: 10.2478/hukin-2014-0017. eCollection 2014 Mar 27. PMID 25031683
- [Background] Urbaniak GC, Plous S. Research randomizer (Version 4.0) [Internet]. 1997 [cited 2024 Dec 2]. Available from: http://www.randomizer.org